CLINICAL TRIAL: NCT07244510
Title: A Phase II, Multicenter, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity of SCT650C in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Efficacy and Safety of SCT650C in Participants With Moderate to Severe Hidradenitis Suppurativa
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT650C-D201
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCT650C high dose Group /Group 1 (Active Comparator): Induction: SCT650C high dose s.c., multiple doses at specified intervals Maintenance: SCT650C high dose s.c., multiple doses at specified intervals
  Interventions: Drug: SCT650C
- SCT650C low dose Group /Group 2 (Active Comparator): Induction: SCT650C low dose s.c., multiple doses at specified intervals Maintenance: SCT650C low dose s.c., multiple doses at special intervels
  Interventions: Drug: SCT650C
- Placebo Group /Group 3 (Placebo Comparator): Induction: Placebo s.c., multiple doses at specified intervals Maintenance: SCT650C high or low dose s.c., multiple doses at specified intervals
  Interventions: Drug: SCT650C

INTERVENTIONS:
Drug: SCT650C — Administered SC
  Other Names: Recombinant anti-IL-17A antibody

SUMMARY:
The purpose of this study is to assess efficacy, safety, pharmacokinetics and immunogenicity of subcutaneous SCT650C in patients with Moderate to Severe Hidradenitis Suppurativa

DETAILED DESCRIPTION:
This is a Phase II, multicenter, double-blinded, placebo-controlled study to evaluate the safety and efficacy of SCT650C in adult participants with Moderate to Severe Hidradenitis Suppurativa. This study includes 3 periods (Screening period, Loading period and Maintenance period ), and ≤ 60 participants in 3 groups (Group 1, 2 and 3)

ELIGIBILITY:
Inclusion Criteria:

1. The participants must be at least 18 years of age at the time of signing the ICF.
2. Study participants must have a diagnosis of HS based on clinical history and physical examination for at least 6 months prior to the baseline visit; diagnosis must be verifiable through medical notes and documentation.
3. Study participants must have HS lesions in at least 2 distinct anatomic areas (eg, left and right axilla), 1 of which must be at least Hurley Stage II or Hurley Stage III at both the Screening and Baseline visits.
4. Study participants must have moderate to severe HS defined as a total of ≥ 5 inflammatory lesions (ie, number of abscesses plus number of inflammatory nodules) at both the Screening and Baseline visits.
5. Study participants must have had a history of inadequate response, intolerance or contraindication to a course of systemic antibiotics for treatment of HS at the Screening Visit as assessed by the investigator.
6. Participants agree to daily use of topical antiseptics on the areas affected by HS lesions while on study treatment. Allowable antiseptic washes are limited to one of the following: chlorhexidine gluconate, benzoyl peroxide, benzalkonium chloride, benzethonium chloride, or dilute bleach in bath water.
7. Participants entering the study while undergoing concomitant treatment with systemic antibiotics (as specified in the protocol) must be on a stable dose. A stable dose is defined as a dosage or regimen that has remained unchanged for at least four weeks prior to baseline and is expected to remain unchanged for at least the first 16 weeks of the study.
8. Female participants must be not of childbearing potential or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception up to 40 weeks after the last administration of the investigational medical product (IMP) and have a negative pregnancy test prior to the first dose. The following methods are considered highly effective when used consistently and correctly:

   1. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable);
   2. combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal);
   3. intrauterine device (IUD);
   4. intrauterine hormone-releasing system (IUS);
   5. bilateral tubal occlusion;
   6. vasectomized partner (where postvasectomy testing had demonstrated sperm clearance);
   7. Sexual abstinence if it is in accordance with a participant's preferred and common lifestyle.

   Note: Participants who use abstinence as a form of birth control must agree to abstain from heterosexual intercourse until 40 weeks after the final dose of IMP. Study personnel must confirm the continued use of abstinence is still in accordance with the participant's lifestyle at regular intervals during the study.

   Male participants with a partner of childbearing potential must be willing to use a condom when sexually active, until 40 weeks after the last administration of IMP.
9. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the participant.

Exclusion Criteria:

1. Study participant has any medical or psychiatric condition could jeopardize or would compromise the study participant's ability to participate in this study as determined by the investigator based on protocol-required assessments.
2. Study participant has a draining fistula count of > 20 at the Baseline Visit.
3. Study participant has any other active skin disease or condition (eg, bacterial cellulitis, candida intertrigo, extensive condyloma) that may, in the opinion of the investigator, interfere with the assessment of HS.
4. Study participant has a diagnosis of sarcoidosis, systemic lupus erythematosus, or active inflammatory bowel disease (IBD).
5. Study participant has a primary immunosuppressive condition, including taking immunosuppressive therapy following an organ transplant or has had a splenectomy.
6. Female study participant who is breastfeeding, pregnant, or plans to become pregnant during the study or within 40 weeks following the final dose of IMP.
7. Study participant has an active infection or history of infection(s) as follows:

   * Any infection requiring systemic treatment within 28 days prior to Baseline;
   * A history of opportunistic, recurrent, or chronic infections that, in the opinion of the investigator, might cause this study to be detrimental to the study participant.

   Opportunistic infections are infections caused by uncommon pathogens (eg, Pneumocystis jirovicii, cryptococcosis), or unusually severe infections caused by common pathogens (eg, cytomegalovirus, herpes zoster).
8. Study participant has any of the following (for more information, refer to Section 9.2):

   * Known active tuberculosis (TB) disease;
   * History of active TB involving any organ system unless adequately treated according to World Health Organization/ Centers for Disease Control and Prevention therapeutic guidance and proven to be fully recovered upon consult with a TB specialist.
   * Latent TB infection (LTBI).
   * High risk of acquiring TB infection.
   * Current or history of NTMB infection.
9. Study participant has an acute or chronic hepatitis B virus, hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection or treponema pallidum antibody (TPPA) positive. Study participants who have evidence of, or tested positive for, hepatitis B or hepatitis C will be excluded.

   1. A positive test for hepatitis B virus is defined as: 1) positive for hepatitis B surface antigen (HBsAg+), or 2) HBsAg is negative, HBcAb is positive and HBV-DNA test results ≥ the upper limit of the reference value of each center or need antiviral treatment.
   2. A positive test for HCV is defined as: 1) positive for hepatitis C antibody (HCVAb+); and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction).
10. Study participants with concurrent malignancy are excluded. Study participants with a history of malignancy within the past 5 years prior to the Screening Visit are excluded, EXCEPT if the malignancy was a cutaneous squamous or basal cell carcinoma, or in situ cervical cancer that has been treated and is considered cured.
11. Study participant has a history of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease.
12. Study participant has had major surgery within the 3 months prior to the Baseline Visit, or has planned major surgery after entering the study.
13. Study participant has any systemic disease (ie, cardiovascular, neurological, renal, liver, metabolic, gastrointestinal, hematological, immunological, etc.) considered by the investigator to be uncontrolled, unstable, or likely to progress to a clinically significant degree during the course of the study.
14. Study participant has had a myocardial infarction or stroke within the 6 months prior to the Screening Visit.
15. Study participant has a history of chronic alcohol or drug abuse within 6 months prior to Screening as evaluated by the investigator based on medical history and interview.
16. Study participant has a history of depression and/or suicidal thoughts or behaviors are considered not suitable for participation in the clinical study by the investigator.
17. The participant has a known hypersensitivity to any excipients of SCT650C.
18. Study participants with prior exposure to biologic agents that block IL-12/23 (e.g., ustekinumab), IL-23 (e.g., risankizumab, guselkumab), or IL-17 (e.g., secukinumab) within 3 months prior to the Baseline visit.
19. Study participants with prior exposure to anti-TNF therapy (e.g., adalimumab, infliximab) for any indication within 2 months prior to the Baseline visit.
20. Study participants who have had prior exposure to other immunomodulatory biologic therapies, including anti-IL-1 (e.g., anakinra, canakinumab), within 3 months or 5 half-lives, whichever is longer, prior to the Baseline visit.
21. Previous treatment with any cell-depleting therapies, including but not limited to anti-CD20 (e.g., rituximab) within 12 months prior to the Baseline visit or until B cell count returns to normal level.
22. Use of traditional medicines or herbal remedies within 28 days prior to the Baseline visit.
23. Study participants have received non-allowable topical therapies (including topical antibiotics) for the treatment of HS within 14 days prior to the Baseline visit.
24. Study participants have received systemic non-biologic therapies (e.g. methotrexate (MTX), cyclosporine A, retinoids, apremilast, phototherapy) for the treatment of HS within 28 days prior to the Baseline visit.
25. For HS and non-HS related pain, participants have received oral concomitant analgesics (including opioids) within 14 days prior to the Baseline visit.

    Exception: Participants may continue on non-opioid analgesics provided that the dose and dosing regimen have been stable for at least 14 days preceding the Baseline visit and are expected to remain stable at least until Week 16 visit.
26. Study participants have received any live vaccine within 8 weeks prior to the first dose of study drug (Baseline), or expect the need for live vaccination during study participation including within 40 weeks after the last dose of study drug administration.
27. Study participants have been treated with any other investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study.
28. Study participant has laboratory abnormalities at Screening, including any of the following:

    * >2× the upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP)
    * Total Bilirubin >2×ULN
    * White blood cell count <3.00×103/μL
    * Absolute neutrophil count <1.5×103/μL
    * Lymphocyte count <500 cells/μL
    * Hemoglobin <8.5g/dL
    * Creatinine >1.5 ×ULN Note: Tests that result in ALT, AST, ALP or total bilirubin up to 25% above the exclusion limit may be repeated for confirmation during the Screening Period. Upon retesting, participants whose ALT, AST, or ALP remain over the above-defined thresholds should not be randomized.
29. Study participant has an estimated glomerular filtration rate (GFR) as measured by Chronic Kidney Disease Epidemiology Collaboration <60mL/min/1.73m2 [GFR (male)=(140-age)ⅹWeight/serum creatinineⅹ1.23; GFR (female)=(140-age)ⅹWeight/serum creatinineⅹ1.04].
30. Study participant has any other laboratory abnormality that, in the investigator's opinion, will prevent the study participant from completing the study or will interfere with the interpretation of the study results.
31. The participant is a SinoCellTech (SCT) employee or is an employee of third-party organizations involved in the study.
32. The participant and/or his or her immediate family member is an employee, volunteer, or other worker at the investigative site, either affiliated or not affiliated with this study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-18 (Estimated); Primary Completion 2027-03-12 (Estimated); Study Completion 2028-02-16 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants achieving HiSCR75 (a 75% reduction from baseline of Hidradenitis Suppurativa Clinical Response [HiSCR]) at Week 16 | Week 16
  HiSCR75 is defined as at least a 75 percent (%) reduction from Baseline in the total abscess and inflammatory nodule (AN) count, with no increase from Baseline in abscess or draining fistula count.

SECONDARY OUTCOMES:
The percentage of participants achieving HiSCR50, HiSCR90, and HiSCR100 at specified time points | Week 48
  HiSCR50 is defined as at least a 50% reduction from Baseline in the total AN count, with no increase from Baseline in abscess or draining fistulas count.
  HiSCR90 is defined as at least a 90% reduction from Baseline in the total AN count, with no increase from Baseline in abscess or draining fistulas count.
  HiSCR100 is defined as at least a 100% reduction from Baseline in the total AN count, with no increase from Baseline in abscess or draining fistulas count.
The percentage of participants achieving HiSCR75 at specified time points | Week 48
  HiSCR70 is defined as at least a 75% reduction from Baseline in the total AN count, with no increase from Baseline in abscess or draining fistulas count.
The percentage of participants who experience ≥ 1 disease flare at specified time points | Week 48
  Flare is defined as a greater than or equal to (>=) 25% increase in AN count with an absolute increase in AN count of >= 2 relative to Baseline.
The change from baseline in the HS-Physician's Global Assessment (HSPGA) at specified time points | Week 48
  The HSPGA is a validated 6-point scale that is used to measure improvement in inflammatory nodules, abscesses, and draining fistulas. This assessment [clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5)] is derived based on totals across all affected body regions.
The change from baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) at specified time points | Week 48
  The IHS4 is a validated tool to dynamically assess HS severity to be used both in real-life and the clinical trials setting. This IHS4 score is calculated as follows: (number of inflammatory nodules multiplied by 1) + (number of abscesses multiplied by 2) + (number of draining fistulae multiplied by 4). A score of 3 or less signifies mild HS, a score of 4-10 signifies moderate HS and a score of 11 or higher signifies severe HS.
The proportion of participants achieving 30% or more reduction in PGA of Skin Pain Numeric Rating Scale (NRS30) at worst among participants with baseline NRS ≥ 3 at specified time points | Week 48
  The PGA of Skin Pain-NRS in the past 24 hours will be used to assess pain "at its worst" due to HS in the last 24 hours. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The PGA of Skin Pain-NRS will be completed by the participant using the Diary.
  NRS30 is defined as at least 30% reduction and at least 1 unit reduction from baseline in Patient's Global Assessment of Skin Pain.
The change from baseline in Dermatology Life Quality Index (DLQI) Total Score at specified time points | Week 48
  The DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life (HRQoL) in adult participants with skin diseases such as eczema, psoriasis, acne, and viral warts. The measure is selfadministered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. The recall period is the last week, and the instrument requires 1 to 2 minutes for completion. Each item has four response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions. Scores range from 0 to 30, with higher scores indicating greater HRQoL, impairment.
Treatment-emergent adverse events (TEAEs), treatment related adverse events (TRAEs), serious adverse events (SAEs) and other safety indicators | Week 48
  A SAE is defined as any untoward medical occurrence that, at any dose: Results in death; Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent disability/incapacity; Is a congenital anomaly/birth defect; Important medical events. TEAEs are defined as those AEs that have a start date on or following the first dose of study treatment.
The drug concentrations of SCT650C at different time points in serum | Week 48
Anti-drug antibodies (ADAs) and neutralizing antibodies (NAbs) | Week 48